CLINICAL TRIAL: NCT04624945
Title: DetectIon of Severe Sepsis In PATients With Neurological haemorrhagE (The DISSIPATE Study)
Acronym: DISSIPATE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Sysmex Asia Pacific (Industry)
Responsible Party: Sponsor
Other Study IDs: 2020/00020
Record Dates: First submitted 2020-11-05; First posted 2020-11-12 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-06

CONDITIONS: Sepsis; Hemorrhage Brain
Keywords: Severe sepsis in patients with neurological haemorrhage
MeSH Terms: conditions — Sepsis; Intracranial Hemorrhages

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SICU cohort: 150 subjects with the admission diagnosis of neurological haemorrhage (e.g. subarachnoid haemorrhage, intracerebral haemorrhage etc), admitted to SICU of National University Hospital, Singapore, who are expected to stay for more than 48 hours, will be recruited and enrolled. Frequency of blood sampling will be stipulated atday 1/2/3/4/5 to draw clinical relevance. An additional 0.5 tablespoonful (7.7ml) of blood will be taken daily from each subject as well as residual blood from routine laboratory test blood samples.
  Interventions: Diagnostic Test: APTT CWA (Activated partial thromboplastin time clot waveform analysis), Procalcitonin and Serological/Inflammatory markers (KL-6, SPA, MIG, Presepsin)

INTERVENTIONS:
Diagnostic Test: APTT CWA (Activated partial thromboplastin time clot waveform analysis), Procalcitonin and Serological/Inflammatory markers (KL-6, SPA, MIG, Presepsin) — Primary Aim: To validate the use of APTT CWA (Activated partial thromboplastin time clot waveform analysis) and ICIS (Intensive Care Infection Score), as early sepsis markers for neurosurgical ICU patients suffering subarachnoid haemorrhage, traumatic brain injury and other intracranial haemorrhages.
  Secondary Aim: To examine the evolution of CWA, immuno-parameters (KL-6, SP-A, MIG, presepsin) and various WBC (white blood cell count) activation markers over the time in relation to diagnosis of sepsis, development of positive blood cultures and mortality or recovery. Blood parameter measurements using a 3-part and 5-part differential analyser will be performed. KL-6, SP-A, MIG, presepsin are serum biomarkers - MIG (Monokine induced by gamma interferon), SP-A (Surfactant protein A), KL-6 (Krebs von den Lungen 6).

SUMMARY:
The research study is to explore novel early predictors and validation of laboratory parameters in the management of sepsis in critically ill patients especially with brain injuries and systemic inflammatory response syndrome (SIRS).

DETAILED DESCRIPTION:
This is a prospective observational study. 150 subjects with the admission diagnosis of neurological haemorrhage (e.g. subarachnoid haemorrhage, intracerebral haemorrhage etc), admitted to SICU of National University Hospital, Singapore, who are expected to stay for more than 48 hours, will be recruited and enrolled. No adverse events are expected as a result of this study as patients do not deviate from the current standard of care. Frequency of blood sampling will be stipulated at day 1/2/3/4/5 to draw clinical relevance. An additional 0.5 tablespoonful (7.7ml) of blood will be taken daily from each subject as well as residual blood from routine laboratory test blood samples. In total, an additional volume of 2.5 tablespoonful (38.5ml) of blood will be collected from each subject over a period of 5 days. Residual blood refers to any leftover blood samples collected for routine laboratory tests which will be shared and used to carry out additional blood tests. All ICU patients will have arterial lines inserted as part of routine care, so there will not be pain from the blood sampling. In the current study, measurements will be made on the routine laboratory haematology, coagulation and immunoassay analyzers. Research blood parameters that are not usually reported as indicated in the background section will be used for the correlation and association analysis to sepsis. In addition, the study team will also be collecting clinical and demographic data of recruited subjects from medical records for purposes of this study.

ELIGIBILITY:
Inclusion Criteria:

* Adults 21 years and above
* Clinical/radiological suspicion or confirmation of neurological haemorrhage

Exclusion Criteria:

* Age below 21 years
* Prisoners
* Known pregnancy
* Do-not-attempt resuscitation status
* Requirement for immediate surgery
* Active chemotherapy/neutropenia (Neutrophil count <1.0 x 109/L)
* Immuno-compromised
* Haematological malignancy
* Treating physician deems aggressive care unsuitable
* Unable to provide informed consent or comply with study requirements

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a prospective observational study. 150 subjects with the admission diagnosis of neurological haemorrhage (e.g. subarachnoid haemorrhage, intracerebral haemorrhage etc), admitted to SICU of National University Hospital, Singapore, who are expected to stay for more than 48 hours, will be recruited and enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-11-25 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
To validate the use of APTT CWA and ICIS, as early sepsis markers for neurosurgical ICU patients suffering subarachnoid haemorrhage, traumatic brain injury and other intracranial haemorrhages. | SICU stay from day 1 to day 5 through to 2 years of blood test completion
  Activated Partial Thromboplastin Time (APTT) clot waveform analysis (CWA) by flow cytometry-based method

SECONDARY OUTCOMES:
To examine the evolution of CWA, immuno-parameters (KL-6, SP-A, MIG, presepsin) and various WBC activation markers over the time in relation to diagnosis of sepsis, development of positive blood cultures and mortality or recovery. | SICU stay from day 1 to day 5 through to 2 years of blood test completion
  Blood parameter measurements using a 3-part and 5-part differential analyser will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Will NH Loh, MBBS, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Scaravilli V, Tinchero G, Citerio G; Participants in the International Multi-Disciplinary Consensus Conference on the Critical Care Management of Subarachnoid Hemorrhage. Fever management in SAH. Neurocrit Care. 2011 Sep;15(2):287-94. doi: 10.1007/s12028-011-9588-6. PMID 21755388
- [Background] Pierrakos C, Vincent JL. Sepsis biomarkers: a review. Crit Care. 2010;14(1):R15. doi: 10.1186/cc8872. Epub 2010 Feb 9. PMID 20144219
- [Background] Jang JH, Park WB, Lim YS, Choi JY, Cho JS, Woo JH, Choi WS, Yang HJ, Hyun SY. Combination of S100B and procalcitonin improves prognostic performance compared to either alone in patients with cardiac arrest: A prospective observational study. Medicine (Baltimore). 2019 Feb;98(6):e14496. doi: 10.1097/MD.0000000000014496. PMID 30732223
- [Background] Pelinka LE, Petto H, Kroepfl A, Schmidhammer R, Redl HJEJoT. Serum Procalcitonin and S100B Are Associated with Mortality after Traumatic Brain Injury. European Journal of Trauma 2003; 29(5): 316-323.
- [Background] Seymour CW, Liu VX, Iwashyna TJ, Brunkhorst FM, Rea TD, Scherag A, Rubenfeld G, Kahn JM, Shankar-Hari M, Singer M, Deutschman CS, Escobar GJ, Angus DC. Assessment of Clinical Criteria for Sepsis: For the Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):762-74. doi: 10.1001/jama.2016.0288. PMID 26903335
- [Background] Chopin N, Floccard B, Sobas F, Illinger J, Boselli E, Benatir F, Levrat A, Guillaume C, Crozon J, Negrier C, Allaouchiche B. Activated partial thromboplastin time waveform analysis: a new tool to detect infection? Crit Care Med. 2006 Jun;34(6):1654-60. doi: 10.1097/01.CCM.0000217471.12799.1C. PMID 16607236
- [Background] Sevenet PO, Depasse F. Clot waveform analysis: Where do we stand in 2017? Int J Lab Hematol. 2017 Dec;39(6):561-568. doi: 10.1111/ijlh.12724. Epub 2017 Sep 6. PMID 28876509
- [Background] Zakariah AN, Cozzi SM, Van Nuffelen M, Clausi CM, Pradier O, Vincent JL. Combination of biphasic transmittance waveform with blood procalcitonin levels for diagnosis of sepsis in acutely ill patients. Crit Care Med. 2008 May;36(5):1507-12. doi: 10.1097/CCM.0b013e3181709f19. PMID 18434897
- [Background] Toh CH, Ticknor LO, Downey C, Giles AR, Paton RC, Wenstone R. Early identification of sepsis and mortality risks through simple, rapid clot-waveform analysis. Implications of lipoprotein-complexed C reactive protein formation. Intensive Care Med. 2003 Jan;29(1):55-61. doi: 10.1007/s00134-002-1557-2. Epub 2002 Nov 22. PMID 12528023
- [Background] Linssen J, Aderhold S, Nierhaus A, Frings D, Kaltschmidt C, Zanker K. Automation and validation of a rapid method to assess neutrophil and monocyte activation by routine fluorescence flow cytometry in vitro. Cytometry B Clin Cytom. 2008 Sep;74(5):295-309. doi: 10.1002/cyto.b.20422. PMID 18431775
- [Background] Weimann K, Zimmermann M, Spies CD, Wernecke KD, Vicherek O, Nachtigall I, Tafelski S, Weimann A. Intensive Care Infection Score--A new approach to distinguish between infectious and noninfectious processes in intensive care and medicosurgical patients. J Int Med Res. 2015 Jun;43(3):435-51. doi: 10.1177/0300060514557711. Epub 2015 Apr 7. PMID 25850686

DOCUMENTS (1):
  • Study Protocol (2020-05-14): https://cdn.clinicaltrials.gov/large-docs/45/NCT04624945/Prot_000.pdf